CLINICAL TRIAL: NCT02338180
Title: A Randomized Clinical Trial on Preventive and Therapeutic Proximal Sealants
Brief Title: Preventive and Therapeutic Proximal Sealants
Acronym: PTPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, CRISTIAN BASILI, DDS, PhD, Associate Professor, Universidad de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Project DIPUV 30/2007
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Dental Caries
Keywords: dental caries; risk assessment; approximal sealant; permanent molar; preventive dentistry; adolescent
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group A (No Intervention): Children with no caries lesion on adjacent surfaces of second primary molar and first permanent molar
- Group B Preventive sealant (Experimental): Children with active caries lesion on distal surfaces of second primary molar and sound mesial surface of first permanent molar. In every children a split mouth design was applied, in one mesial surfaces of first molar randomize selected received a proximal preventive sealants, and the other remain as a control
  Interventions: Other: proximal preventive sealants
- Group C Therapeutic sealant (Experimental): Children with active caries lesion on distal surfaces of second primary molar and active lesion on mesial surface of first permanent molar. In every children a split mouth design was applied, in one mesial surfaces of first molar randomize selected received proximal therapeutic sealant, and the other remain as a control
  Interventions: Other: proximal preventive sealants; Other: proximal therapeutic sealant

INTERVENTIONS:
Other: proximal preventive sealants — On sound mesial surfaces of first permanent molars adjacent to a caries active lesion of second primary molar, after 4-6 days with an orthodontic separating rubber ring around the approximal contact area. The test site was isolated with cotton rolls or a rubber dam. The surface of 6m was etched with 35% phosphoric acid for 20 sec, washed with water and then air-dried. The sealant (Concise Sealant; 3M ESPE) was applied and light-cured for 20 sec each on the occlusal, buccal and lingual sides. After polymerization, the sealant was inspected for complete coverage.
  Other Names: Concise Sealant (3M ESPE)
  Arms: Group B Preventive sealant; Group C Therapeutic sealant
Other: proximal therapeutic sealant — On mesial surfaces of first permanent molars with caries active lesion adjacent to a caries active lesion of second primary molar , after 4-6 days with an orthodontic separating rubber ring around the approximal contact area. The test site was isolated with cotton rolls or a rubber dam. The surface of 6m was etched with 35% phosphoric acid for 20 sec, washed with water and then air-dried. The sealant (Concise Sealant; 3M ESPE) was applied and light-cured for 20 sec each on the occlusal, buccal and lingual sides. After polymerization, the sealant was inspected for complete coverage.
  Other Names: Concise Sealant (3M ESPE)
  Arms: Group C Therapeutic sealant

SUMMARY:
It is of clinical importance to arrest the development of approximal caries at an early stage. The potential for initial caries to develop into manifest lesions has motivated studies on the use of sealants to arrest the progression of caries on both occlusal and approximal tooth surfaces.

Therefore, the aim of the present study was to follow-up and examine after 3.5 years, the efficacy of sealing caries-free or non-cavitated mesial surfaces of first permanent molars abutting lesions on the distal surfaces of second primary molars. The null hypothesis tested here was that preventive and therapeutic sealants do not prevent the development or slow the progression of dental caries over a period of 3.5 years in comparison to non-sealed control surfaces.

DETAILED DESCRIPTION:
The study population comprised 121 schoolchildren aged 8 to 10 years in a high-caries community in Valparaiso, Chile. They were examined clinically and radiographically, divided into 3 groups, and treated accordingly: children in Group A had no carious lesions on the approximal surfaces of 05d-6m and received no sealants; those in group B had active caries on 05d and received a preventive sealant on the caries-free 6m; and those in group C had active caries on 05d with an initial active lesion on 6m and received a therapeutic sealant on 6m. After 3.5 years, standardized follow-up radiographs were obtained for the children that remained.

ELIGIBILITY:
Inclusion Criteria:

* children with high rate of caries in the primary dentition
* active caries on the distal surfaces of the second primary molars at least on both sides of the mouth
* children with no lesions on the adjacent tooth surfaces on the second primary and first permanent molars were included as a general control group

Exclusion Criteria:

* children using medication containing sucrose or with a negative effect on salivary flow
* children using orthodontic devices
* children who refuses to participate

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 390 (Actual)
Dates: Start 2009-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of active lesion developed on first molar mesial surfaces | 3.5 years (42-44 months)
  Outcome will be measured by a radiographical examination (standardized posterior bitewings) 3.5 years after the preventive or therapeutical proximal sealants have been applied.

CONTACTS AND LOCATIONS:
Overall Officials: Cristian P Basili, DDS, PHD, Principal Investigator — University of Valparaiso
Locations (1):
- Dental Reference Center Simon Bolivar, Viña del Mar, Región de Valparaíso, Chile

REFERENCES:
- [Background] Martignon S, Ekstrand KR, Gomez J, Lara JS, Cortes A. Infiltrating/sealing proximal caries lesions: a 3-year randomized clinical trial. J Dent Res. 2012 Mar;91(3):288-92. doi: 10.1177/0022034511435328. Epub 2012 Jan 17. PMID 22257664
- [Result] Ammari MM, Soviero VM, da Silva Fidalgo TK, Lenzi M, Ferreira DM, Mattos CT, de Souza IP, Maia LC. Is non-cavitated proximal lesion sealing an effective method for caries control in primary and permanent teeth? A systematic review and meta-analysis. J Dent. 2014 Oct;42(10):1217-27. doi: 10.1016/j.jdent.2014.07.015. Epub 2014 Jul 24. PMID 25066832
- [Result] Gomez SS, Basili CP, Emilson CG. A 2-year clinical evaluation of sealed noncavitated approximal posterior carious lesions in adolescents. Clin Oral Investig. 2005 Dec;9(4):239-43. doi: 10.1007/s00784-005-0010-7. Epub 2005 Sep 16. PMID 16167153